CLINICAL TRIAL: NCT03801733
Title: A Phase 1, Three-Part, Open-label Study in Healthy Adult Volunteers to Assess Vadadustat as a Perpetrator in Drug-Drug Interactions With Rosuvastatin, Sulfasalazine, Pravastatin, Atorvastatin and Simvastatin
Brief Title: Drug-Drug Interaction Study of Vadadustat With Rosuvastatin, Sulfasalazine, Pravastatin, Atorvastatin and Simvastatin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Akebia Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: AKB 6548 CI 0030
Record Dates: First submitted 2018-12-27; First posted 2019-01-11 (Actual); Last update posted 2019-03-22 (Actual); Status verified 2019-03

CONDITIONS: Drug Interaction Potentiation
Keywords: Vadadustat; Normal Healthy volunteers; Pharmacokinetics; Rosuvastatin; Sulfasalazine; Pravastatin; Atrovastatin; Simvastatin
MeSH Terms: interventions — vadadustat; Simvastatin; Rosuvastatin Calcium; Atorvastatin; Pravastatin; Sulfasalazine

STUDY DESIGN:
Intervention Model Description: This is a three-part sequential design study. Part 2 will be initiated based upon the outcome of Part 1 and Part 3 will be initiated after completion of Part 2.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Rosuvastatin, Vadadustat (Experimental): Part 1: Subjects will receive rosuvastatin 20 mg alone, vadadustat 600 mg alone, followed by rosuvastatin 20 mg in combination with vadadustat 600 mg in a fixed-sequence dosing design.
  Interventions: Drug: Vadadustat; Drug: Rosuvastatin
- Sulfasalazine. Pravastatin, Vadadustat (Experimental): Part 2, Arm 1: Subjects will receive sulfasalazine 500 mg alone followed by sulfasalazine 500 mg in combination with vadadustat 600 mg once a day in a fixed-sequence dosing design.
  Part 2, Arm 2: Subjects will receive pravastatin 40 mg alone followed by pravastatin 40 mg in combination with vadadustat 600 mg once a day in a fixed-sequence dosing design.
  Interventions: Drug: Vadadustat; Drug: Pravastatin; Drug: Sulfasalazine
- Atorvastatin, Simvastatin, Vadadustat (Experimental): Part 3, Arm 1: Subjects will receive atorvastatin 40 mg alone followed by atorvastatin 40 mg in combination with vadadustat 600 mg once a day in a fixed-sequence dosing design.
  Part 3, Arm 2: 24 subjects will receive simvastatin 40 mg alone followed by simvastatin 40 mg in combination with vadadustat 600 mg once a day in a fixed-sequence dosing design.
  Interventions: Drug: Vadadustat; Drug: Simvastatin; Drug: Atorvastatin

INTERVENTIONS:
Drug: Vadadustat — Oral dose of 600 mg QD
  Other Names: AKB 6548
Drug: Simvastatin — Oral Simvastatin
  Arms: Atorvastatin, Simvastatin, Vadadustat
Drug: Rosuvastatin — Oral Rosuvastatin
  Arms: Rosuvastatin, Vadadustat
Drug: Atorvastatin — Oral Atorvastatin
  Arms: Atorvastatin, Simvastatin, Vadadustat
Drug: Pravastatin — Oral Pravastatin
  Arms: Sulfasalazine. Pravastatin, Vadadustat
Drug: Sulfasalazine — Oral Sulfasalazine
  Arms: Sulfasalazine. Pravastatin, Vadadustat

SUMMARY:
This is a Phase 1, three-part, open-label study to evaluate vadadustat as a perpetrator in drug-drug interactions with rosuvastatin, sulfasalazine, pravastatin, atorvastatin and simvastatin in healthy male and female subjects.

DETAILED DESCRIPTION:
This is a Phase 1, three-part, open-label study to evaluate vadadustat as a perpetrator in drug-drug interactions with rosuvastatin, sulfasalazine, pravastatin, atorvastatin, and simvastatin in healthy male and female subjects. Thirty-four (34) subjects will be enrolled in Part 1 (rosuvastatin) and based on review of the PK and safety/tolerability data, a decision will be made on whether to proceed with Part 2. Part 2 consists of 2 arms (sulfasalazine and pravastatin). Twenty-six (26) subjects will be enrolled into each arm. Part 3 consists of 2 arms (atorvastatin and simvastatin). Twenty-four (24) subjects will be enrolled into each arm after enrollment in Part 2 is completed. Subjects will be in the study for up to 72 days, including a 28-day screening period, 6-14 day in clinic period, and a 30-day follow up period post last dose. Blood samples for PK analysis will be collected at pre-defined time points throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Male or female between 18 and 55 years of age, inclusive, at time of informed consent
* Body mass index between 18.0 and 30.0 kg/m2, with a minimum body weight of 45 kg for females and 50 kg for males, inclusive.

Exclusion Criteria:

* Current or past clinically significant history of cardiovascular, cerebrovascular, pulmonary, gastrointestinal, hematologic, renal, hepatic, immunologic, metabolic, urologic, neurologic, dermatologic, psychiatric, or other major disease. History of cancer (except treated non-melanoma skin cancer) or history of chemotherapy use within 5 years prior to Screening; History of latent or active tuberculosis (TB).
* Positive test results for human immunodeficiency virus (HIV) antibody; 12. Positive test results of hepatitis B surface antigen (HBsAg), or positive hepatitis C virus antibody (HCVab) within 3 months prior to screening, or positive test results for human immunodeficiency virus antibody (HIVab) at Screening
* Taking any prescription medication or over the counter multi-vitamin supplement, or any non-prescription products (including herbal-containing preparations but excluding acetaminophen) within 14 days prior to Day -1.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 134 (Actual)
Dates: Start 2018-06-17 (Actual); Primary Completion 2018-11-24 (Actual); Study Completion 2018-11-24 (Actual)

PRIMARY OUTCOMES:
Area under plasma concentration-time curve from time 0 to last quantifiable concentration (AUClast) of rosuvastatin, sulfasalazine, pravastatin and simvastatin | Up to 10 weeks
Area under plasma concentration-time curve from time 0 to infinity (AUCinf) of rosuvastatin, sulfasalazine, pravastatin and simvastatin | Up to 10 weeks
Maximum observed plasma concentration (Cmax) of rosuvastatin. sulfasalazine, pravastatin, atorvastatin and simvastatin | Up to 10 weeks
Area under plasma concentration-time curve (AUCtau) of atorvastatin | Up to 10 weeks

SECONDARY OUTCOMES:
Time to maximum observed plasma concentration (Tmax) of rosuvastatin, sulfasalazine, pravastatin, atorvastatin, and simvastatin | Up to 10 weeks
Elimination rate constant (Kel) of rosuvastatin, sulfasalazine, pravastatin, atorvastatin, and simvastatin | Up to 10 weeks
Terminal half-life (t½) of rosuvastatin, sulfasalazine, pravastatin, atorvastatin, and simvastatin | Up to 10 weeks
Apparent total body clearance (CL/F) of rosuvastatin, sulfasalazine, pravastatin, atorvastatin, and simvastatin | Up to 10 weeks
Percentage of extrapolated area under the curve from time t to infinity (%AUCextrap or Residual Area) of rosuvastatin, sulfasalazine, pravastatin, atorvastatin, and simvastatin | Up to 10 weeks
Area under plasma concentration-time curve from time 0 to last quantifiable concentration (AUClast) of sulfasalazine metabolites, sulfapyridine and 5-ASA (mesalamine | Up to 10 weeks
Area under plasma concentration-time curve from time 0 to infinity (AUCinf) of sulfasalazine metabolites, sulfapyridine and 5-ASA (mesalamine | Up to 10 weeks
Maximum observed plasma concentration (Cmax) of sulfasalazine metabolites, sulfapyridine and 5-ASA (mesalamine | Up to 10 weeks
Time to maximum observed plasma concentration (Tmax) of sulfasalazine metabolites, sulfapyridine and 5-ASA (mesalamine | Up to 10 weeks
Elimination rate constant (Kel) of sulfasalazine metabolites, sulfapyridine and 5-ASA (mesalamine | Up to 10 weeks
Terminal half-life (t½) of sulfasalazine metabolites, sulfapyridine and 5-ASA (mesalamine | Up to 10 weeks
Area under the plasma concentration-time curve for a dosing interval (AUCtau) of atorvastatin metabolites, o-hydroxyatorvastatin; p-hydroxyatorvastatin | Up to 10 weeks
Maximum observed plasma concentration (Cmax) of atorvastatin metabolites, o-hydroxyatorvastatin; p-hydroxyatorvastatin | Up to 10 weeks
Time to maximum observed plasma concentration (Tmax) of atorvastatin metabolites, o-hydroxyatorvastatin; p-hydroxyatorvastatin | Up to 10 weeks
Area under plasma concentration-time curve from time 0 to last quantifiable concentration (AUClast) of simvastatin metabolite | Up to 10 weeks
Area under plasma concentration-time curve from time 0 to infinity (AUCinf) of simvastatin metabolite | Up to 10 weeks
Maximum observed plasma concentration (Cmax) of simvastatin metabolite | Up to 10 weeks
Time to maximum observed plasma concentration (Tmax) of simvastatin metabolite | Up to 10 weeks
Elimination rate constant (Kel) of simvastatin metabolite | Up to 10 weeks
Terminal half-life (t½), of simvastatin metabolite | Up to 10 weeks
Reporting of treatment emergent adverse events (TEAE) as reported by the study subjects | Up to 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Akebia Inc, Study Director — Akebia Therapeutics
Locations (1):
- InVentiv Health Clinique Inc., Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided